CLINICAL TRIAL: NCT04598165
Title: Mobile WACh NEO Randomized Clinical Trial: Mobile Phone 2-Way Short Message Service (SMS) Versus Control to Reduce Neonatal Mortality in Kenya
Brief Title: Mobile WACh NEO: Mobile Solutions for Neonatal Health and Maternal Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Kenyatta National Hospital (Other Government)
Responsible Party: Principal Investigator, Jennifer Unger, Associate Professor, Department of Obstetrics and Gynecology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006395; 1R01HD098105-01 (NIH)
Record Dates: First submitted 2020-10-02; First posted 2020-10-22 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Neonatal Death; Perinatal Death; Depression
Keywords: SMS; mHealth; neonate; mortality; depression; Kenya
MeSH Terms: conditions — Perinatal Death; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1) Interactive two-way SMS dialogue or 2) Control (no SMS), using 1:1 allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive two-way SMS dialogue (Experimental): Participants will receive automated SMS messages with prompts to reply. They will have the ability to both respond to and initiate SMS dialogue. Trained Study Nurses will monitor and respond to participant messages.
  Interventions: Behavioral: Interactive two-way SMS dialogue
- No SMS Control (No Intervention): Control receiving standard of care.

INTERVENTIONS:
Behavioral: Interactive two-way SMS dialogue — We will utilize Mobile WACh, a human-computer hybrid system that enables seamless two-way SMS communication and patient tracking, to provide consistent support to women and their infants during the peripartum period and 6 weeks into the baby's life. Women will receive automated theoretically grounded SMS messages targeting the appropriate peripartum period and will have the capability to respond and spontaneously message a nurse based at the clinic. During pregnancy, automated SMS will be delivered weekly. Two weeks prior to the participant's estimated due date (EDD), daily messaging will begin, and will continue for two weeks after delivery is ascertained. Thereafter, SMS will be delivered every other day for the remaining four weeks. Women who experience pregnancy or infant loss will be enrolled into an infant loss track where they will receive messages of support.
  Arms: Interactive two-way SMS dialogue

SUMMARY:
To improve neonatal mortality, it is critical to engage families, especially mothers, in essential newborn care (ENC) and appropriate care-seeking for neonatal illness as well as to support maternal mental health and self-efficacy. This randomized controlled trial (RCT) aims to determine the effect and mechanisms of a two- way mobile health (mHealth) SMS intervention, Mobile WACh NEO, on neonatal mortality, essential newborn practices, care-seeking and maternal mental health at four sites in Kenya.

DETAILED DESCRIPTION:
High-impact essential newborn care practices and interventions are available to support neonatal survival, but coverage remains a challenge in sub-Saharan Africa, where neonatal mortality is unacceptably high. Many newborns continue to die at home without health care services being sought. The reasons are multifactorial, at the societal, health system, and family levels. Decisions made within the household and the family's ability to reach care play a large part in determining neonatal outcomes. It is estimated that up to 80% of neonatal and child deaths may have delays in recognition of infant illness and decision to seek care. Two-way mobile health (mHealth) communication strategies can enable mothers to remotely interact with a healthcare worker (HCW) and receive real-time education, counseling, encouragement, motivation and decisional guidance to support care-seeking decisions and ultimately neonatal health and survival.

The investigators developed a unique two-way SMS platform (Mobile WACh) that combines automated SMS messaging and dialogue with a HCW. The team adapted this approach for intensive neonatal support and evaluations (Mobile WACh NEO). Mobile WACh NEO (MWN) enhances the benefits of SMS messaging by engaging mothers with SMS communication and bringing timely information and support - asking critical questions at crucial times in order to assess the needs and health of newborns and assist in care seeking decisions.

This is a randomized controlled trial of the MWN intervention among 5,020 participants (2,510 MWN arm, 2,510 control arm) to determine the effect of MWN on neonatal mortality, essential newborn care, care seeking, and maternal mental health in the first 6 weeks postpartum.

Aim 1: To determine the effect of Mobile WACh NEO on neonatal mortality, compared to no SMS control.

Aim 2: To examine the effect of Mobile WACh NEO on maternal implementation of essential newborn care and care seeking behavior.

Aim 3: To examine the effects of Mobile WACh NEO on maternal social support, self-efficacy and depression.

Finally, investigators will explore the associations between maternal mental health, implementation of essential newborn care, neonatal care seeking and participant engagement by SMS.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* 28-36 weeks gestation
* Daily access to a mobile phone (own or shared) on the Safaricom network
* Willing to receive SMS
* Able to read and respond to text messages in English, Kiswahili or Luo, or have someone in the household who can help

Exclusion Criteria:

* Currently enrolled in another research study
* Previous participant in the Mobile WACh NEO RCT (i.e. with a new pregnancy)

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5020 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Unger, MD, MPH, Principal Investigator — Brown University; John Kinuthia, MBChB, MMed, Study Director — Kenyatta National Hospital
Locations (6):
- Kenya (6):
  - Ahero Sub-District Hospital, Ahero, Kisumu County
  - Bondo Sub-County Referral Hospital, Bondo
  - Rachuonyo County Hospital, Homa Bay
  - Kisumu County Hospital, Kisumu
  - Mathare North Health Centre, Nairobi
  - Riruta Health Center, Nairobi

IPD SHARING:
Plan to Share IPD: Yes
Data from Mobile WACh NEO will be available at end of the project by contacting the study team at the University of Washington (neor01@uw.edu).
Time Frame: At the end of the project.

REFERENCES:
- [Background] Ronen K, Choo EM, Wandika B, Udren JI, Osborn L, Kithao P, Hedstrom AB, Masinde M, Kumar M, Wamalwa DC, Richardson BA, Kinuthia J, Unger JA. Evaluation of a two-way SMS messaging strategy to reduce neonatal mortality: rationale, design and methods of the Mobile WACh NEO randomised controlled trial in Kenya. BMJ Open. 2021 Dec 23;11(12):e056062. doi: 10.1136/bmjopen-2021-056062. PMID 34949631
- [Derived] Unger JA, Kinuthia J, Wandika B, Hedstrom A, Wetzler E, Udren JI, Masinde M, Choo EM, Schultes O, Kithao P, Moraa J, Akinyi E, Osborn L, Nzove E, Richardson BA, Kumar M, Wamalwa D, Ronen K. The impact of interactive text communication on neonatal mortality in Kenya: a randomized controlled trial. Nat Med. 2025 Jun;31(6):1847-1854. doi: 10.1038/s41591-025-03576-z. Epub 2025 Mar 12. PMID 40075230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women were recruited when attending routine antenatal care through referral to study staff. Those interested were asked to provide verbal consent for screening to assess eligibility, and if eligible, they were invited to participate in the study. Women were followed until 6 weeks postpartum but their infants were not considered enrolled. Infant outcomes were obtained from the participants and considered participant outcomes.
Groups:
- Interactive Two-way Text Messaging Dialogue: Participants will receive automated SMS messages with prompts to reply. They will have the ability to both respond to and initiate SMS dialogue. Trained Study Nurses will monitor and respond to participant messages.
  Interactive two-way SMS dialogue: We will utilize Mobile WACh, a human-computer hybrid system that enables seamless two-way SMS communication and patient tracking, to provide consistent support to women and their infants during the peripartum period and 6 weeks into the baby's life. Women will receive automated theoretically grounded SMS messages targeting the appropriate peripartum period and will have the capability to respond and spontaneously message a nurse based at the clinic. During pregnancy, automated SMS will be delivered weekly. Two weeks prior to the participant's estimated due date (EDD), daily messaging will begin, and will continue for two weeks after delivery is ascertained. Thereafter, SMS will be delivered every other day for the remaining four weeks. Women who experience pregnancy or infant loss will be enrolled into an infant loss track where they will receive messages of support.
Period: Completed 6-week Follow-up
Arm/Group | Interactive Two-way Text Messaging Dialogue | No SMS Control
Started | 2509 | 2511
Completed | 2471 | 2470
Not Completed | 38 | 41
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 26 | 33
Not completed — Ineligible | 4 | 3
Not completed — Partner refusal | 0 | 1
Period: Included in Intention to Treat Analysis
Arm/Group | Interactive Two-way Text Messaging Dialogue | No SMS Control
Started | 2509 (Participants did not need to complete the 6-week visit in order to contribute to the primary ITT neonatal mortality analysis as the death could have been reported prior to this visit.) | 2511 (Participants did not need to complete the 6-week visit in order to contribute to the primary ITT neonatal mortality analysis as the death could have been reported prior to this visit.)
Completed | 2442 | 2442
Not Completed | 67 | 69
Not completed — Ineligible for inclusion in analysis | 67 | 69

BASELINE CHARACTERISTICS:
Population: Seven (7) enrolled participants excluded from analysis due to ineligibility.
Groups:
- Total: Total of all reporting groups
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control | Total
Number analyzed (Participants) | 2505 | 2508 | 5013
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [22 to 29] | 25 [22 to 29] | 25 [22 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2505 | 2508 | 5013
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2505 | 2508 | 5013
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 2505 | 2508 | 5013
<12 years of education [Count of Participants; unit: Participants] | 1037 | 1005 | 2042
Household crowding (>3 people per room) [Count of Participants; unit: Participants] | 399 | 371 | 770
Married/cohabitating [Count of Participants; unit: Participants] | 2000 | 2050 | 4050
Employed [Count of Participants; unit: Participants] | 943 | 921 | 1864
Shares mobile phone [Count of Participants; unit: Participants] | 299 | 240 | 539
Can read SMS unassisted [Count of Participants; unit: Participants] | 2500 | 2501 | 5001
Can write SMS unassisted [Count of Participants; unit: Participants] | 2492 | 2501 | 4993
Received health SMS messages from another program [Count of Participants; unit: Participants] | 635 | 577 | 1212
Intimate partner violence in last month [Count of Participants; unit: Participants] | 91 | 98 | 189
Primigravida [Count of Participants; unit: Participants] | 864 | 828 | 1692
Twins [Count of Participants; unit: Participants] | 42 | 39 | 81
Estimated gestational age in weeks at baseline [Mean (Inter-Quartile Range); unit: weeks] | 31.6 [29.9 to 33.7] | 31.4 [29.7 to 33.7] | 31.6 [29.7 to 33.7]
HIV positive [Count of Participants; unit: Participants] | 218 | 208 | 426
Elevated depressive symptoms defined as a score ≥13 on Edinburgh Postnatal Depression Score (EPDS) [Count of Participants; unit: Participants] | 78 | 81 | 159
Self-reported social support score using the MOS social support survey [Median (Inter-Quartile Range); unit: units on a scale from 0-100] — Higher numbers indicate more social support.
  units on a scale from 0-100 | 80.3 [65.8 to 100] | 82.9 [65.8 to 100] | 81.6 [65.8 to 100]
Parenting self-efficacy using the Karitane Parenting Confidence Scale (KPCS) [Median (Inter-Quartile Range); unit: units on a scale from 0-45] — Higher numbers indicate more confidence.
  units on a scale from 0-45 | 45 [41 to 45] | 45 [41 to 45] | 45 [41 to 45]
Enrollment clinic [Count of Participants; unit: Participants]
  Facility 1 | 185 | 184 | 369
  Facility 2 | 480 | 481 | 961
  Facility 3 | 197 | 197 | 394
  Facility 4 | 766 | 772 | 1538
  Facility 5 | 458 | 459 | 917
  Facility 6 | 419 | 415 | 834

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Mortality
Description: Death during 1st 28 days of life
Time Frame: 28 days postpartum
Population: Intention-to-treat for participants with a known infant outcome at 6 weeks postpartum. Seventy-two (72) participants excluded from the Overall Number of Participants Analyzed, due to stillbirth.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2442 | 2442
Participants | 46 | 37
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; We estimated a sample size of 5000 to detect a risk ratio of ≤0.53 assuming a neonatal mortality rate of 23 per 1000 in the control arm with 80% power and, 95% confidence and taking into account a 10% attrition. Multiple imputation with chain equations (MICE) was used to impute missing values for any outcome with greater than 10% missingness. Any variables associated with the outcome or outcome missingness were included in the imputation model; Test type: Superiority; p = 0.314, Poisson regression — The primary intention to treat analysis was adjusted for differences in exposure to other SMS programs and phone ownership. The threshold for statistical significance was p=0.05; Risk Ratio (RR) = 1.25, 95% CI 2-sided [0.81 to 1.92] — SMS group is the numerator

2. Secondary Outcome: Early Neonatal Mortality
Description: Death during 1st 7 days of life
Time Frame: 7 days postpartum
Population: Intention-to-treat for participants with a known infant outcome at the 7th day of life. Seventy-two (72) stillbirths were removed from analysis cohort. This includes 13 participants for whom an outcome is not known at 6 weeks of life for the primary outcome. Seventy-two (72) stillbirths were removed from analysis cohort.Seventy-two (72) participants excluded from the Overall Number of Participants Analyzed, due to stillbirth.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2450 | 2447
Participants | 38 | 28
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.217, Poisson regression — The intention to treat analysis was adjusted for differences in exposure to other SMS programs and phone ownership. We corrected for multiple comparisons using the Benjamini-Hochberg method. The threshold for statistical significance was p=0.05; Risk Ratio (RR) = 1.36, 95% CI 2-sided [0.84 to 2.21] — SMS group is the numerator

3. Secondary Outcome: Initiation of Early Breastfeeding
Description: Number of participants initiating breastfeeding in 1st hour of life
Time Frame: 1 hour postpartum
Population: This population includes participants who did not experience a stillbirth or infant death by 2 weeks postpartum, who attended the 2 week follow-up visit, who did not decline to answer and those for whom data was not missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2088 | 2007
Participants | 1510 | 1402
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; We estimated a sample size of 5000 to detect a risk ratio of ≤0.53 assuming a neonatal mortality rate of 23 per 1000 in the control arm with 80% power and, 95% confidence and assuming 10% attrition. With this sample size, assuming alpha=0.0045 (Bonferroni adjusted for 11 tests), we also had 80% power to detect a risk ratio of 1.05 in early initiation of breast feeding assuming 80% uptake in controls; Test type: Superiority; p = 0.064, Poisson regression — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.04, 95% CI 2-sided [1.00 to 1.08] — SMS group is the numerator

4. Secondary Outcome: Exclusive Breastfeeding
Description: Exclusive breastfeeding at 6-week visit
Time Frame: 6-weeks postpartum
Population: This population includes participants who did not experience a stillbirth or infant death by 6 weeks postpartum, who attended the 6 week follow-up visit, who did not decline to answer and those for whom data was not missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2386 | 2396
Participants | 2190 | 2217
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; We estimated a sample size of 5000 to detect a risk ratio of ≤0.53 assuming a neonatal mortality rate of 23 per 1000 in the control arm with 80% power and, 95% confidence and assuming 10% attrition. With this sample size, assuming alpha=0.0045 (Bonferroni adjusted for 11 tests), we also had 80% power to detect a risk ratio of 1.05 in exclusive breast feeding assuming 80% uptake in controls; Test type: Superiority; p = 0.363, Poisson regression — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.98 to 1.01] — SMS group is the numerator

5. Secondary Outcome: Thermal Care
Description: Number of participants not giving infant a bath in 1st 24 hours of life
Time Frame: 24 hours postpartum
Population: This population includes participants who did not experience a stillbirth or infant death by 2 weeks postpartum, whose infants did not die on the first day of life, who did not decline to answer and those for whom data was not missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2332 | 2343
Participants | 2245 | 2232
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; We estimated a sample size of 5000 to detect a risk ratio of ≤0.53 assuming a neonatal mortality rate of 23 per 1000 in the control arm with 80% power and, 95% confidence and assuming 10% attrition. With this sample size, assuming alpha=0.0045 (Bonferroni adjusted for 11 tests), we also had 80% power to detect a risk ratio of 1.11 in application of substances to the cord or delaying first bath assuming 50% in controls; Test type: Superiority; p = 0.093, Poisson regression — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.01, 95% CI 2-sided [1.00 to 1.02] — SMS group is the numerator

6. Secondary Outcome: Cord Care
Description: Number of participants with no application of substances to cord
Time Frame: 2-weeks postpartum
Population: This population includes participants who did not experience a stillbirth or infant death by 2 weeks postpartum, those who did not decline to answer and those for whom data was not missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2374 | 2378
Participants | 1123 | 1104
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.353, Poisson regression — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.97 to 1.09] — SMS group is the numerator

7. Secondary Outcome: Home Provision of Kangaroo Mother Care
Description: Number of participants providing any duration of skin-to-skin care on ≥10 of the first 14 days at home, among low birthweight or preterm infants
Time Frame: 14 days at home postpartum
Population: Only among preterm and/or low birth weight live births.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 185 | 174
Participants | 12 | 10
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; We estimated a sample size of 5000 to detect a risk ratio of ≤0.53 assuming a neonatal mortality rate of 23 per 1000 in the control arm with 80% power and, 95% confidence and assuming 10% attrition. With this sample size, assuming alpha=0.0045 (Bonferroni adjusted for 11 tests), we also had 80% power to detect a risk ratio of 1.53 in provision of Kangaroo Mother Care assuming 25% in controls; Test type: Superiority; p = 0.751, Poisson regression — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.50 to 2.61] — SMS group is the numerator

8. Secondary Outcome: Maternal Knowledge of Neonatal Danger Signs
Description: Number of danger signs or symptoms successfully named
Time Frame: Up to 6-weeks postpartum
Population: For this time-varying outcome, data for the 6-week visit are presented here. This population includes those who did not decline to answer and those for whom data was not missing. Data are missing for those experienced an infant loss by the 6-week visit.
Measure: Median (Inter-Quartile Range); unit: Number of danger signs named
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2389 | 2397
Number of danger signs named | 3 [2 to 4] | 2 [2 to 3]
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; We estimated a sample size of 5000 to detect a risk ratio of ≤0.53 assuming a neonatal mortality rate of 23 per 1000 in the control arm with 80% power and, 95% confidence and assuming 10% attrition. With this sample size, assuming alpha=0.0045 (Bonferroni adjusted for 11 tests), we also had 80% power to detect a risk ratio of 1.04 in number of danger signs correctly named assuming median of 3 in controls; Test type: Superiority; p = 0.431, Poisson generalized estimating equations — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.00, 95% CI 2-sided [1.00 to 1.01] — n (%) are values at 6-week visit, and RR compares change over time for enrollment, 2- and 6-week visits. SMS group is the numerator

9. Secondary Outcome: Appropriate Care-seeking
Description: Proportion of illness episodes with danger signs in which the clinic was attended and/or where the infant was hospitalized irrespective of danger signs reported in 1st 18 weeks of life (study follow-up period).
Time Frame: 18 weeks postpartum
Population: Only in infants with illness episodes with danger signs and/or where the infant was hospitalized irrespective of danger signs reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 214 | 172
Participants | 204 | 160
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; We estimated a sample size of 5000 to detect a risk ratio of ≤0.53 assuming a neonatal mortality rate of 23 per 1000 in the control arm with 80% power and, 95% confidence and assuming 10% attrition. With this sample size, assuming alpha=0.0045 (Bonferroni adjusted for 11 tests), we also had 80% power to detect a risk ratio of 1.11 in appropriate care seeking assuming 1 clinic visit in the 6-weeks postpartum for controls; Test type: Superiority; p = 0.321, Poisson regression — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.98 to 1.08] — SMS group is the numerator

10. Secondary Outcome: Elevated Depressive Symptoms
Description: Score above diagnostic threshold (>=13) for Edinburgh Postnatal Depression Scale. Possible scores are 0-30, with a higher score indicating a higher likelihood of possible depressive illness.
Time Frame: Enrollment through 6-weeks postpartum
Population: This population includes participants who attended the 6 week visit, those who did not decline to answer and those for whom data was not missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2467 | 2462
Participants | 38 | 40
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; We estimated a sample size of 5000 to detect a risk ratio of ≤0.53 assuming a neonatal mortality rate of 23 per 1000 in the control arm with 80% power and, 95% confidence and assuming 10% attrition. With this sample size, assuming alpha=0.0045 (Bonferroni adjusted for 11 tests), we also had 80% power to detect a risk ratio of 0.76 in elevated depression symptoms assuming 19% in controls; Test type: Superiority; p = 0.650, Poisson generalized estimating equations — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.98 to 1.04] — [estimate comment as in outcome 8, analysis 1]

11. Secondary Outcome: Social Support
Description: Score using Medical Outcomes Study (MOS) Social Support Survey. Possible scores are 0-100, with a higher score indicating higher levels of social support.
Time Frame: Enrollment through 6-weeks postpartum
Population: For this time-varying outcome, data for the 6-week visit are presented here. This population includes those who did not decline to answer and those for whom data was not missing.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2469 | 2466
score on a scale | 84.2 [69.7 to 100] | 84.2 [68.4 to 100]
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; Test type: Superiority; p = 0.071, Linear generalized estimating equations — [p-value comment as in outcome 2, analysis 1]; Coefficient = 0.09, 95% CI 2-sided [-0.007 to 0.18] — n (%) are values at 6-week visit, and RR compares change over time for enrollment, 2- and 6-week visits. SMS group is the numerator. Coefficient (95% CI) for linear GEE using enrollment, 2- and 6-week visits

12. Secondary Outcome: Self-efficacy
Description: Score using the Karitane Parenting Confidence Scale. Possible scores are 0-45, with higher scores indicating higher levels of parenting confidence.
Time Frame: Enrollment through 6-weeks postpartum
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
Number analyzed (Participants) | 2253 | 2247
score on a scale | 45 [43 to 45] | 45 [43 to 45]
Statistical Analysis 1: Comparison: Interactive Two-way SMS Dialogue vs No SMS Control; Test type: Superiority; p = 0.190, Linear generalized estimating equations — [p-value comment as in outcome 2, analysis 1]; Coefficient = 0.02, 95% CI 2-sided [-0.01 to 0.04] — [estimate comment as in outcome 11, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire span of the study from enrollment through the participants' study exit at 18 weeks postpartum.
Description: Participants (i.e. mothers) were systematically assessed for events throughout their study enrollment; information provided was by their self-report. Adverse events include social harms, encompassing abuse, suicidal behavior, and psychological distress. Serious adverse events include infant hospitalization and death; stillbirth; maternal hospitalization, death, and disappearance.
Arm/Group | Interactive Two-way SMS Dialogue | No SMS Control
All-Cause Mortality (participants affected / at risk) | 2/2505 | 2/2508
Serious Adverse Events (participants affected / at risk) | 171/2505 | 114/2508
Other Adverse Events (participants affected / at risk) | 7/2505 | 2/2508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Interactive Two-way SMS Dialogue (N=2505) | No SMS Control (N=2508)
Maternal death (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Infant death (Pregnancy, puerperium and perinatal conditions) | 54/2441 (55) | 39/2442 (40) — Deaths of live-born infants. Stillbirths and missing outcome data excluded from denominator.
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 34 (34) | 39 (39)
Maternal hospitalization (General disorders) | 33 (35) | 11 (12)
Infant hospitalization (General disorders) | 90/2471 (94) | 46/2469 (46) — Hospitalization of live-born infants. Stillbirths excluded from denominator.
Maternal disappearance (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interactive Two-way SMS Dialogue (N=2505) | No SMS Control (N=2508)
Social harm (Social circumstances) | 7 (7) | 2 (4)

LIMITATIONS AND CAVEATS:
The individual rather than cluster level randomization may have led to contamination. Nurse text responses came mostly during the day and thus limited the intervention's ability to address time-sensitive concerns. Limited access to facility records also posed challenges to understanding details of clinical care. The study was not powered to find a mortality difference between the arms among babies who died after discharge from delivery hospitalization, for whom the intervention was designed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04598165/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT04598165/SAP_001.pdf
  • Informed Consent Form (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT04598165/ICF_002.pdf